CLINICAL TRIAL: NCT07327554
Title: Xmouv - Assessment of the Evolution of Lumbar Spine Movement Fluidity Using Xsens Inertial Sensors in Subjects With Chronic Low Back Pain Before and After Rehabilitation
Brief Title: Assessment of the Evolution of Lumbar Spine Movement Fluidity Using Xsens Inertial Sensors in Subjects With Chronic Low Back Pain Before and After Rehabilitation
Acronym: Xmouv
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL25_0310; 2025-A02160-49 (Other: ID-RCB)
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; kinematic; jerk; instability catch; aberrant movement patterns
MeSH Terms: conditions — Low Back Pain; Fasciculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compare Movement Fluidity Before and After Rehabilitation (Experimental): Evolution of Movement Fluidity Before and After Rehabilitation in patients with chronic low back pain
  Interventions: Device: X-sens sensor

INTERVENTIONS:
Device: X-sens sensor — kinematic movement measurement using 5 Xsens inertial sensors (Awinda) placed on the head, thoracic vertebrae (T8), lumbar vertebrae (L1, L4), and sacrum (S1), before and after the rehabilitation program (ten working days). Movement will be measured during standardized tasks including 3 lumbar spine flexions and 3 right and left lumbar rotations. Movements will be recorded by the sensors at a frequency of 100 Hz.

SUMMARY:
Low back pain, defined as pain located between the thoracolumbar junction and the lower gluteal fold, becomes chronic in 8% of patients. As the leading cause of disability worldwide, it has major individual and medico-economic consequences.

Three-dimensional biomechanical analysis allows exploration of movement alterations related to low back pain. Although several parameters have already been studied (maximum joint range of motion (ROM), lumbopelvic rhythm, movement variability, gait), no consistent kinematic profile has emerged. Movement fluidity, assessed by the presence of jerks (brief movement disturbances), remains under-described despite its relevance in evaluating movement quality.

Invistigators hypothesize that lumbar spine movement fluidity during flexion improves after a rehabilitation program and correlates with clinical response.

This project stands out by exploring a rarely studied parameter (movement fluidity) and integrating it as a potential indicator for rehabilitation monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years inclusive
* BMI between 18-30 kg/m²
* Chronic low back pain lasting more than three months
* Rehabilitation care in the Physical Medicine and Rehabilitation Department of Montpellier University Hospital

Exclusion Criteria:

* Sciatica episode within the last three months
* Traumatic, tumoral, or infectious cause of low back pain
* History of spinal, pelvic, or hip fracture
* Inflammatory rheumatism
* Lumbar arthrodesis
* Severe scoliosis
* Subject with a legal protection measure (guardianship, curatorship)
* Subject under legal protection
* Subject not affiliated to a social security system or not benefiting from such a system
* Absence of informed written consent
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between the evolution of trunk flexion movement fluidity and the evolution of disability before and after rehabilitation program | 2 weeks
  Movement velocity will be measured during flexion using Xsens inertial measurement units (head, T8, L1, L4, S1). Velocity profiles will identify acceleration and deceleration phases. Movement fluidity will be quantified by a normalized jerk metric: the count of local minima and maxima on the angular velocity curve divided by flexion/extension duration (peaks/s). This normalization accounts for variations in movement speed between individuals and measurement sessions, providing a standardized measure of movement smoothness where lower values indicate more fluid motion.
  Disability will be measured by the change in the score of Oswestry Disability Index (ODI) questionary between the first and last day of rehabilitation. The ODI questionary contains ten topics concerning intensity of pain and activities of daily life. Each question is scored on a scale of 0-5 where zero indicates the least amount of disability and 5 indicating most severe disability. The ODI scale range from 0 to 100

SECONDARY OUTCOMES:
Changes in range of motion (ROM) between the first and last day of rehabilitation program | 2 weeks
  The evolution of trunk range of motion (degree) between the first and last day of rehabilitation will be measured during flexion and rotation movement using Xsens inertial measurement units positioned on the head and at T8, L1, L4 and S1. ROM represents the maximal angular displacement reached by the trunk during the movement and allows identification of the contribution of different segments.
Changes in maximum angular velocity between the first and last day of rehabilitation program | 2 weeks
  The evolution of maximum angular velocity (degrees per second) between the first and last day of rehabilitation will be measured during flexion and rotation movements using Xsens inertial measurement units positioned on the head and at T8, L1, L4, S1. Angular velocity reflects the peak speed at which the trunk segment rotates during motion. The movement velocity will be assessed both locally and globally.
Changes in lumbopelvic rhythm between the first and last day of rehabilitation program | 2 weeks
  Changes in lombopelvic rhythm between the first and last day of rehabilitation will be assessed during the flexion using Xsens inertial measurement units positioned on the head and at T8, L1, L4, S1. lombopelvic rhythm represents the coordination and relative contribution of lumbar spine and pelvic motion during bending tasks.
Changes in functional disability between the first and last day of rehabilitation program | 2 weeks
  The evolution of functional disability between the first and last day of rehabilitation program will be measured by the Oswestry Disability Index (ODI) questionary. This self-completed questionnaire contains ten topics concerning intensity of pain, and activities of daily life. Each topic category contains 6 statements describing a growing degree of relative severity to a particular activity. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 where zero indicates the least amount of disability and 5 indicating most severe disability. The ODI scale range from 0 to 100 where zero corresponds
Changes in pain between the first and last day of rehabilitation program | 2 weeks
  The evolution of pain intensity between the first and last day of rehabilitation program will be measured by Visual Analogue Scale (VAS), ranging from 0 to 10, where 0 represents no pain and 10 represents maximum pain.
Changes in psychological impact between the first and last day of rehabilitation program | 2 weeks
  The evolution of psychological impact between the first and last day of rehabilitation program will be measured by the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 7 items designed to evaluate depression and 7 for the anxiety. Each item is rated on a 4-point scale ranging, from 0 = no, not at all, to 3 = yes.
Changes in kinesiophobia between the first and last day of rehabilitation program | 2 weeks
  The evolution of kinesiophobia between the first and last day of rehabilitation program will be measured by the Tampa Scale of Kinesiophobia (TSK) measuring the fear that pain may occur as a result of movement. The TSK is a questionnaire of 17 questions rated by a four-point ordinal scale, ranging, from 1 for strongly disagree, to 4 for strongly agree.
Changes in catastrophizing between the first and last day of rehabilitation program | 2 weeks
  The evolution of catastrophizing between the first and last day of rehabilitation program will be measured by the Pains Catastrophizing Scale (PCS) assessing the extent of catastrophic thinking related to pain. The PCS consists of 13 items, each rated on a 5-point Likert scale (0 = not at all to 4 = all the time).
Changes in fears and beliefs regarding work and physical activity between the first and last day of rehabilitation program | 2 weeks
  The evolution of beliefs related to fear and avoidance of pain between the first and last day of rehabilitation program will be measured by the Fear avoidance Belief Questionnaire (FABQ). The FABQ comprises 16 items. Patients are asked to rate each item on a scale ranging from 0 for 'strongly disagree' to 6 for 'strongly agree'. It consists of two sub-scores: FABQ Physical (FABQ-PA), comprising 5 items and assessing beliefs related to physical activity. FABQ Work (FABQ-W), comprising 11 items and assessing beliefs related to work.
Changes in Schober index between the first and last day of rehabilitation program | 2 weeks
  The Schober index is a clinical assessment tool used to evaluate lumbar spine flexion and mobility. The test is performed with the subject standing upright. The examiner marks a point over the fifth lumbar vertebra (L5) and a second point 10 cm above the first. The subject is then asked to bend forward maximally, and the distance between the two marks is measured again. A normal mobility is characterized by an increase in the distance between the two markers of 4 to 7 cm.
Changes in fingertip-to-floor distance between the first and last day of rehabilitation program | 2 weeks
  The distance between the tips of the fingers and the floor (in cm) is measured when the subject standing with knees straight, leans forward as far as possible in an attempt to touch the floor with their fingers.
Changes in heel-to-buttock distance between the first and last day of rehabilitation program | 2 weeks
  The distance between the heel and the buttock (in cm) is measured when the subject lying in a prone position. The examiner performs passive flexion of the knee by bringing the heel closer to the buttock and measures the distance
Changes in popliteal angle between the first and last day of rehabilitation program | 2 weeks
  The popliteal angle (in degree) is measured between the axis of the leg and the axis of the hip when the subject is lying supine and the examiner performs passive flexion of the hip to 90° followed by passive extension of the knee. The measurement is taken on both sides.
Changes in Sorensen test between the first and last day of rehabilitation program | 2 weeks
  The Sorensen Test is a clinical assessment used to measure the isometric endurance of the trunk muscles. The subject lies prone on a table with the upper edge of the iliac crest aligned with the table edge, and the lower body secured with straps at the pelvis, knees, and ankles. With arms crossed over the chest, the subject maintains the upper body in a horizontal position unsupported.
  The test duration is recorded (in seconds) until the subject can no longer hold the position.
Changes in Shirado test between the first and last day of rehabilitation program | 2 weeks
  The Shirado Test is a clinical assessment used to measure the strength and endurance of the abdominal muscles. The subject lies in a supine position with hips and knees flexed at 90 degrees, and arms crossed over the chest. The position is timed (in seconds) and the subject is asked to hold it for as long as possible. The test ends when the subject is no longer able to maintain the position.
Changes in isometric endurance of trunk muscles between the first and last day of rehabilitation program | 2 weeks
  The isometric endurance of trunk muscles is assessed by the ratio between the time taken in the Shirado test (in seconds) and the time taken in the Sorensen test (in seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Isabel TAVARES, MD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided